CLINICAL TRIAL: NCT03983707
Title: A Multicentre Prospective Observational Study to Evaluate the Utilisation, Effectiveness and Safety of Purastat® in the Management of Gastrointestinal Bleeding
Brief Title: A Evaluation of the Utilisation, Effectiveness and Safety of Purastat® in the Management of Gastrointestinal Bleeding
Acronym: POPS
Status: Completed | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Collaborators: 3-D Matrix Europe SAS (Industry); Gloucestershire Hospitals NHS Foundation Trust (Other); Cambridge University Hospitals NHS Foundation Trust (Other); University Hospital Birmingham NHS Foundation Trust (Other); Nottingham University Hospitals NHS Trust (Other); Mid and South Essex NHS Foundation Trust (Other); East Kent Hospitals University NHS Foundation Trust (Other Government); University College London Hospitals (Other); North Tees and Hartlepool NHS Foundation Trust (Other); Brighton and Sussex University Hospitals NHS Trust (Other); King's College Hospital NHS Trust (Other); Imperial College Healthcare NHS Trust (Other); Heart of England NHS Foundation Trust (Unknown); The Leeds Teaching Hospitals NHS Trust (Other); Barts & The London NHS Trust (Other); London North West Healthcare NHS Trust (Other); Manchester University NHS Foundation Trust (Other Government); Oxford University Hospitals NHS Trust (Other); Glasgow Royal Infirmary (Other); Guy's and St Thomas' NHS Foundation Trust (Other); Northern Care Alliance NHS Foundation Trust (Other); University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: PHT/2018/39
Record Dates: First submitted 2019-04-23; First posted 2019-06-12 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2022-09

CONDITIONS: Gastrointestinal Bleeding; Delayed Bleeding
Keywords: Purastat
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Purastat® — Use of Purastat®

SUMMARY:
Problem statement

GI bleeding can arise from peptic ulcers, malignancy, angiodysplasia or during endoscopic resection procedures such as endoscopic mucosal resection and endoscopic submucosal dissection. This is conventionally treated using heat therapy or clips. These methods carry a risk of thermal injury or perforation. Purastat® is a novel synthetic haemostatic agent licensed as a CE marked device for use in GI bleeding. It also has the potential to enhance endoscopic mucosal wound healing and may play a role in preventing delayed bleeding. However, clinical data on its effectiveness in the GI tract is limited. Prospective data collection on the range of indications for Purastat® use and outcome data related to clinical effectiveness, safety and feasibility is required to inform clinicians about the best use for this agent.

Research question / hypothesis

To establish a prospective registry study to collect outcome data related to the use of Purastat® for the clinical management of GI bleeding or prevention of bleeding

Study Design

Prospective multicentre cohort study

Study Participants

Adults with GI bleeding or a high risk of bleeding during endoscopic procedures where Purastat® has been used

Follow-up duration

All patients will be followed up as per standard clinical care where applicable

Planned Study Period

2 years

Primary Objective

To assess the effectiveness of Purastat® as a haemostatic agent when used in the treatment of GI bleeding

Secondary Objectives

To assess the incidence of delayed bleeding after use of Purastat®, defined as procedure related bleeding up to 28 days following endoscopic resection To evaluate the rate of rebleeding following primary application of Purastat® for haemostasis To assess the technical feasibility and ease of use of Purastat® when used in the treatment or prevention of GI bleeding To monitor any unexpected reactions that may be attributed to the use of Purastat® To describe utilisation patterns in different clinical centres (indication, patient characteristics etc) and to observe trends in utilisation over time

DETAILED DESCRIPTION:
Problem statement

GI bleeding can arise from peptic ulcers, malignancy, angiodysplasia or during endoscopic resection procedures such as endoscopic mucosal resection and endoscopic submucosal dissection. This is conventionally treated using heat therapy or clips. These methods carry a risk of thermal injury or perforation. Purastat® is a novel synthetic haemostatic agent licensed as a CE marked device for use in GI bleeding. It also has the potential to enhance endoscopic mucosal wound healing and may play a role in preventing delayed bleeding. However, clinical data on its effectiveness in the GI tract is limited. Prospective data collection on the range of indications for Purastat® use and outcome data related to clinical effectiveness, safety and feasibility is required to inform clinicians about the best use for this agent.

Research question / hypothesis

To establish a prospective registry study to collect outcome data related to the use of Purastat® for the clinical management of GI bleeding or prevention of bleeding

Study Design

Prospective multicentre cohort study

Study Participants

Adults with GI bleeding or a high risk of bleeding during endoscopic procedures where Purastat® has been used

Follow-up duration

All patients will be followed up as per standard clinical care where applicable

Planned Study Period

2 years

Primary Objective

To assess the effectiveness of Purastat® as a haemostatic agent when used in the treatment of GI bleeding

Secondary Objectives

To assess the incidence of delayed bleeding after use of Purastat®, defined as procedure related bleeding up to 28 days following endoscopic resection To evaluate the rate of rebleeding following primary application of Purastat® for haemostasis To assess the technical feasibility and ease of use of Purastat® when used in the treatment or prevention of GI bleeding To monitor any unexpected reactions that may be attributed to the use of Purastat® To describe utilisation patterns in different clinical centres (indication, patient characteristics etc) and to observe trends in utilisation over time

ELIGIBILITY:
Inclusion Criteria:

* Active GI bleeding or high risk for active GI bleeding

Exclusion Criteria:

* Variceal or arterial bleeding

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults with GI bleeding or a high risk of bleeding during endoscopic procedures where Purastat® is used
Sampling Method: Non-Probability Sample
Enrollment: 379 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Effectiveness of Purastat® in controlling bleeding | Day 1 (intraprocedural bleeding)
  Number (and proportion) of bleeds successfully controlled by application of Purastat®
Effectiveness of Purastat® in controlling bleeding | Day 28 (delayed bleeding)
  Number (and proportion) of bleeds successfully controlled by application of Purastat®

SECONDARY OUTCOMES:
Effectiveness of Purastat® in preventing delayed bleeding | Day 28
  Delayed bleeding rate
Technical feasibility of use of Purastat® | Day 1 (periprocedural)
  Any difficulty in Purastat application (yes/no)
Unexpected reactions that may be attributed to the use of Purastat® | Day 28
  Occurrence of Suspected Unexpected Serious Adverse Reactions (SUSAR) related to Purastat®
Patterns of Purastat® usage | 24 months
  Purastat® utilisation (including indications)

CONTACTS AND LOCATIONS:
Overall Officials: Pradeep Bhandari, Principal Investigator — Portsmouth Hospitals NHS Trust
Locations (1):
- Queen Alexandra Hospital, Portsmouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No